CLINICAL TRIAL: NCT04271852
Title: An Experimental Protocol for the Study of Brain Functional Magnetic Resonance Imaging in Female With Urgent Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2019-09-112
Record Dates: First submitted 2019-11-28; First posted 2020-02-17 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Urinary Incontinence, Urge
MeSH Terms: conditions — Urinary Incontinence, Urge

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UUI patients (Experimental): 50 UUI patients will have biofeedback treatment once a week.
  Interventions: Device: bio-feedback treatment
- Control (No Intervention)

INTERVENTIONS:
Device: bio-feedback treatment — 50 patients will treated with phenix u2 and phenix u4 treating equipment。
  Arms: UUI patients

SUMMARY:
Background: Patients' life quality and physical and mental health are seriously affected by Urgent Urinary Incontinence(UUI). The cause is not clear at present. It has been found that the injury of the prefrontal lobe and damage to the surrounding cerebral cortex leads to significant lower urinary tract dysfunction. Therefore, some scholars believe that urinary axis of the brain exist between the urinary system and the central nervous system, and the two are controlled by each other. Therefore, to study central conduction in patients with UUI and changes of physiology, pathology, brain chemical, brain structure in brain functional area caused by central sensitivity, in particular, changes in urine control cognition and midbrain limbic system (including memory function areas) in the brain, is beneficial to more in-depth understanding of its pathogenesis and treatment options. The Functional Magnetic Resonance Imaging provides a possibility for the study.

Method / design:Taking female UUI patients as target, through questionnaire survey, voiding diary, specialist physique, examination,ultrasonic examination of pelvic floor muscle, urodynamic examination and three sequence magnetic resonance scanning, after analyzing structural image of brian, resting functional images, dispersion tensor image, comparing with the normal control group and the female UUI group, before and after behavioral therapy in patients with UUI, and those who have no urinary incontinence and those who still have urinary incontinence after behavioral treatment, specific brain function biomarkers for female UUI patients are found and the brain function mechanism of the female UUI is to be explored in this project.

Discussion: This study breaks through the traditional limitations on the cause of incontinence.And it is the first time,the mental/behavior indicators of uui patients were combined with fMRI(Functional Magnetic Resonance Imaging) to explore biomarkers of brain and brain structural changes in patients .Then,it is becoming more and more important that the personalized treatment by building a UUI digital model using fMRI.

DETAILED DESCRIPTION:
The study is a randomized controlled trial that study on the mechanism of brain function in women with urgent urinary incontinence by using fMRI. According to the exclusion criteria, 50 healthy volunteers and 50 UUI patients are recruited to carry out the related experimental research.This study had been approved by the Ethics Committee of the second affiliated Hospital of Wenzhou Medical University (No. LCK2019-291) .

1.50 UUI patients and 50 healthy volunteers who meet the inclusion criteria were selected.

(1) Approved by the Scientific Research Ethics Review Committee of the second affiliated Hospital of Wenzhou Medical University, 20- 70 years old female volunteers are recruited by studying advertising, reminding volunteers that the study is recruiting women with well bladder control function through the answer to the relevant questionnaires as a screening tool.

2.1 Healthy volunteers (n=50) should empty thier bladder first ；than they perform a fMRI scan.

2.2 The selected patients (n=50) will be inserted into 8F catheter for urine emptying, determination of bladder pressure and injection of aseptic water. First of all, the subjects empty their urine through the catheter, perform a fMRI scan first, and perform the following cycle module after the first scan is complete:①Paused for 11s ②.Injecting 22ml aquae sterilisata into bladder through catheter (completed in 11s ) ③.Paused for 11s ④.withdraw15ml liquid through catheter (completed in 11s ) , running 1-5 modules in circles until the subject issues a urination signal. With the subject's consent, the above cycle is repeated once, to exclude dropout who will be marked as a failure in the study. The rest of the patients completed the above circulation and patients with urine leakage scan the fMRI again.

3.Every fMRI scan of each subject included in the study will be scanned on GE-Discovery 7503T magnetic resonance machine for three sequences (T1,rsfMRI, DTI). The total scanning time is about 25 minutes. The brain structural image (T1) uses GE BRAVO sequence for about 5 minutes and the specific parameters are as follows:TR/TE=7.7/3.4 ms, Flip angle=12°, FOV=256 mm×256 mm, Resolution=256×256, Slice per volume=176, Slice thickness=1 mm. The rsfMRI(resting-state functional magnetic resonance) uses a single EPI sequence for about 10 minutes and the specific parameters are as follows.TR/TE=2000/30 ms, Flip angle=90°, FOV=220 mm×220 mm, Resolution=64×64, Slice thickness=4 mm, Slices per volume=32, Number of volumes=230. The diffusion tensor image (DTI) uses a single diffusion-weighted spin echo EPI sequence for about 10 minutes and the specific parameters are as follows:TR/TE=8000/80 ms, Flip angle=90°, FOV=256 mm×256 mm, Resolution=128×128, Slice thickness=2 mm, Slices per volume=75. In order to use the latest method to analyze the gray microstructure of the brain,investigators will choose two non-zero b values:b=1000 s/mm2 , with a total of 23 dispersion directions; b = 2000 s/mm2 , with a total of 49 dispersion directions.

4. The 50 UUI patients who completed the above trial will be treated with behavioral therapy for 3 months under the guidance of medical staff. The behavioral therapy includes: (1) changes in the way of life including quit smoking, lose weight, keep a normal bowel movement, drinking water in a regular basis, no coffee and white spirit, don't eat spicy and irritating foods, regular urination and defecation, etc. (2) Bladder training: set a urination schedule, with a short interval of time at first, when feeling urination is urgent, the tension of bladder can be alleviated by slow deep breathing and mental transfer to increase the interval of urination gradually. (3) have pelvic floor muscle exercise by drawing up the anus such as, hold on to exhaust and defecate from the anus. The contraction lasts 3, 5 or 10 seconds. And then completely relax the anus. The relaxation time is equal to the drawing up time of anus with 10 to 15 times per exercise, and3 to 5 times a day.

5.Patients with UUI who completed 3 months' behavioral therapy repeat the above 2 -5 study steps again.

6.Relevant research parameters:Image parameters of brain function:investigators will first get the whole brain voxel image parameters and investigators get local gray matter density in structural image. Local degree will be gotten in functional image while local fractional anisotropy, FA will be gotten in the dispersion tensor image. Then by calculating global gray matter density, global degree and global FA, investigators will get the global variables of the brain function (structural, functional and white matter connection anisotropy) of the participants.

7. Data analysis:①By comparing the image parameters of whole brain function with those of the normal control group (Student t-test group comparison, two tails, p < 0.05/3=0.017 （family-wise correction）),investigators will verify one of research assumptions, that is, whether the brain of the UUI patient has a significant change in function and structure (structural, functional, and white matter connection anisotropy) as compared to the brain of a normal person; At the same time, By comparing the image parameters of whole brain voxel image parameters with those of the normal control group (student t group comparison，two tails, p < 0.05, cluster size > 30 (cluster-wise correction)), investigators find out those specific significantly altered data (questionnaire for quality of life of urinary incontinence I-QOL, FSFI- female sexual function index assessment) that shows significant linear correlation (Pearson Correlation, p <0.05, with age as covariate) with praxiology where the brain region is a unique biomarker of brain function in patients with UUI. ②UUI patients will be divided into two groups after treatment, that is, the symptoms of urinary incontinence disappeared after treatment (abbreviated as the disappeared) and the urinary incontinence was not relieved after treatment (abbreviated as the the unrelieved). Through comparing the image parameters (F-test one-way ANOVA，two tails, p < 0.05/3=0.017 (family-wise correction))，of whole brain function among the three groups (normal control group, the disappeared group and unrelieved group), investigators will verify the second hypothesis, that is, for patients with UUI whose symptoms of urinary incontinence disappear after behavioral therapy, whether the function and structure of the brain (structural, functional and white matter connectivity) will change reversibly and return to its original state;

③ Through analysis of changes in behavioral data before and after treatment (questionnaire for quality of life of urinary incontinence I-QOL, FSFI- female sexual function index assessment) and linear correlation analysis of all-brain functional image parameters (Pearson Correlation, p < 0.05, age as covariate), investigators can verify the third hypothesis, that is, the degree of unrelieved urinary incontinence after UUI behavior therapy is significantly correlated with his / her brain function and structural changes.

8.Data analysis tools:FSL software will be applied for brain function image analysis, and MATLAB and SPSS for data statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* People in the group should meet the following inclusion criteria:

  * 20-70 years old, medical history ≥ 3 months.
  * According to International Continence Society, ICS, people in the group should be patients diagnosed with UUI.

Exclusion Criteria:

* Exclusion standards should be met by both patient group and the control group ( Not included in if meeting one of the following items ):

  * Scan contraindication ：（1）reactive metal.(2)cardiac pacemaker.(3)magnetic implantation.(3)no spring steel wire in eyelid.(4)artificial cochlea.(5)electrodes/wires, pregnancy, etc.
  * Patients with severe organ diseases ：·（1）liver disease.(2)lung disease.(3)kidney disease.(4)Other diseases that may interfere with the effectiveness and safety assessment of the test or may place the patient at some particular risk.
  * People who is unable to cooperate with each other.
  * A neurological or other medical disease that affects the function of the central nervous system ：（1） anemia.（2） vitamin B12 deficiency .（3）folic acid deficiency.
  * People who abuse drug.
  * People who has dependence history
  * Hyperthyroidism in active period
  * cerebrovascular disease (e.g. transient ischemic attack, ischemic or hemorrhagic stroke, aneurysm)
  * Central nervous system infection
  * Alcoholic dementia
  * Uncontrolled epilepsy
  * Autoimmune disease
  * Diabetes mellitus
  * Detrusor hyperreflexia (cystitis, tuberculosis, tumor, stone, bladder outlet obstruction) and other organic lesion.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Femal
Enrollment: 100 (Estimated)
Dates: Start 2019-10-23 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessing change of the number of leakages was used to assess the severity of urinary incontinence. | Baseline,3th month
  By ues of voiding diaries.The more frequent leakage, the more serious incontinence.
  Baseline：
Brain regional gray matter density change of subjects | Baseline,3th month
  All subjects will be scanned by MRI for contrasting anatomic brain image，and the brain regional gray matter density will be calculated from the contrasting anatomical image.
Brain functional connectivity strength | Baseline,3th month
  All the subjects will be scanned by MRI for functional brain images，and the brain functional connectivity strengths will be calculated from the contrasting anatomical images,with number 1presents the maximum positive connectivity between two different brain regions,number-1presents maximum negative connectivity,and number 0 presents 0 connectivity.
  The change of brain connection intensity in three months.

SECONDARY OUTCOMES:
Assessing change of POP-Q measurements were used to assess pelvic floor prolapse. | Baseline,3th month
  POP-Q（Pelvic Organ Prolapse Quantitive examination）：Contrast changes in POP-Q measurements.Measure nine point include Ab，Ba，Ap，Bp,Tvl，gh，pb，C，D.
  POP-Q is based on hymen (0 point), Six points of the anterior wall, posterior wall and the top of the vagina were used as indicator points (two points of the anterior wall, AA and Ba, two points of the posterior wall, AP and BP, two points of the top, C and D), The changes of the six points relative to the hymen were measured in scale (the indication points were negative in the inner side of the hymen margin and positive in the outer side of the hymen margin), and the prolapse was quantified.
  At the same time, total vaginal length (TVL) was recorded, At the same time, the length of gonadal hiatus (GH) was recorded At the same time, the length of perineal body (PB) was recorded. Aa、Ba、Ap、Bp：Normal range at -3cm. C、D：Normal range at -Tvl to-（Tvl-2）
Assessing change of the number of millimeters of rectocele used to evaluate the prolapse of the posterior wall of the vagina. | Baseline,3th month
  （By Urodynamic examination）Measurement of rectocele：Degree of swelling 0-15mm is mild，>15mm or above is severe.
  The degree of rectocele was compared before and after three months.
Assessing change of the number of millimeters of prolapse used to assess the extent of prolapse. | Baseline,3th month
  （By Urodynamic examination）The distance between the uterus and the margin of hymen.The unit is mm.
Assessing change of the measurement of detrusor compliance was used to assist in the evaluation of acute incontinence.（By Urodynamic examination） | Baseline,3th month
  （By Urodynamic examination）Compliance: The ratio of increased detrusor pressure to increased bladder capacity (c = △ v / △ p).(>20ml/cmH2O).Maximum bladder compliance = maximum bladder capacity ÷ (filling resting pressure-empty resting pressure).
  The compliance of bladder was higher than that of three months ago.The unit is >20ml/cmH2O.
Assessing change of Bladder neck mobility, used to assess the presence of stress urinary incontinence. | Baseline,3th month
  Bladder neck activity > 15mm, increased bladder neck activity
Assessing change of the number of millimeters of cystocele used to evaluate the prolapse of the anterior wall of the vagina. | Baseline,3th month
  （By Urodynamic examination）Measurement of cystocele：Degree of swelling 0-10mm is mild，>10mm or above is severe.
  The degree of cystocele was compared before and after three months.

OTHER OUTCOMES:
Positive and negative mood effect of subject | Baseline,3th month
  The positive and negative affect schedule has two mood scales,one measuring positive affect and the other measuring negative affect，The lowest possible score for each question is 1,the highest possible score rror each question is 5.
  Affect Schedule(Sections1,3,5,9,10,12,14,16,17,19)：Score can range from 10 to50，with higher scores representing higher levels of positive affect.
  Negative Affect Schedule(Sections2,4,6,7,8,11,13,15,18,20)，Score can range from 1 to 50，with lower scores representing lower levels of negative affect.
PISQ-12 change of subjects | Baseline,3th month
  Pelvic organ prolapse/Urinary incontinence Sexual questionnaire short from PISQ-12:The PISQ-12 questionnaire have 12 questions，the highest possible score for each question is 4,The lowest possible score for each question is 0,Score can range from 0 to 48.With higher scores representing higher levels of sexual satisfaction.
I-QOL change of subjects | Baseline,3th month
  The Urinary Incontinence-Specific Quality of Life Instrument（I-QOL）：This questionnaire have 22 questions，the highest possible score for each question is 5,The lowest possible score for each question is 0,Final Score is equal to（total score-22）/88*100.Final score can range from 0 to 100.With higher scores representing higher levels of quality of life.
FSFI change of subjects | Baseline,3th month
  The Female Sexual Function Index (FSFI)：This questionnaire have 19 questions.The higher the score, the better the function Score less than 25 points, diagnosed as sexual dysfunction Less than 3.6 points of single item indicates decreased sexual desire or difficulty in sexual arousal, less than 3.9 points indicate difficulty in vaginal lubrication, less than 4 points indicate difficulty in orgasm, and less than 4.4 points indicate decreased sexual satisfaction.
SF-12 change of subjects | Baseline,3th month
  This questionnaire have 12 questions： Sections1,4,5,6,7,8,9,10,11,12：Each question have 5 options.The lowest possible score for each question is 1,the highest possible score for each question is 5.
  Sections2,3：Each question have 2 options,The highest possible score for each question is 5,the lowest possible score for each question is1.
  Total score can range from 12 to 56.With higher scores representing lower levels of life quality.
The severity of depression of subjects | Baseline,3th month
  Beck's Depression index add up the 21 questions.The highest possible score for each question is 3,The lowest possible score for each question is 0,The possible total scores can range from 0 to 63.With the higher value represent a worse depression.
PFID-20 change of subjects | Baseline,3th month
  Pelvic Floor Distress Inventory Questionnaire - Short Form 20 (PFDI-20) ：This questionaire have 3 parts.
  1. POPDI-6:This parts focus on the symptom of pelvic.This part have 6 questions,the highest possible score for each question is 4,The lowest possible score for each question is 0.With the higher value represent a worse pelvic function.
  2. CRADI-8:This parts focus on the symptom of colorectal.This part have 8 questions,the highest possible score for each question is 4,The lowest possible score for each question is 0.With the higher value represent a worse defecation.
  3. UDI-6:This parts focus on the symptom of urinary.This part have 6 questions,the highest possible score for each question is 4,The lowest possible score for each question is 0.With the higher value represent a worse urination.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gynecology of Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China